CLINICAL TRIAL: NCT02040246
Title: Comparison of Metformin and Repaglinide Monotherapy in the Treatment of New Onset Type 2 Diabetes Mellitus in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jing Ma, Consultant, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSFC-81070651
Record Dates: First submitted 2013-12-25; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repaglinide (Experimental): Initial dose of repaglinide 0.5 mg once daily. During the dose titration period of 1 week, the dose of repaglinide could be titrated up to 1 mg three times daily, according to fasting glucose values. The minimal dose was repaglinide 0.5 mg three times daily.
  Interventions: Drug: Repaglinide
- Metformin (Active Comparator): Initial dose of metformin 250mg once daily. During the dose titration period of 1 week, the dose could be titrated up to metformin 500 mg three times daily, according to fasting glucose values.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Repaglinide — Initial dose of repaglinide 0.5 mg once daily. During the dose titration period of 1 week, the dose of repaglinide could be titrated up to 1 mg three times daily, according to fasting glucose values. The minimal dose was repaglinide 0.5 mg three times daily.
  Arms: Repaglinide
Drug: Metformin — Initial dose of metformin 250mg once daily. During the dose titration period of 1 week, the dose could be titrated up to metformin 500 mg three times daily, according to fasting glucose values.
  Arms: Metformin

SUMMARY:
The prevalence of diabetes is up to 11.6% according to the data released in 2013 by the China Noncommunicable Disease Surveillance Group.Less than 40% of all diagnosed-diabetes were well controlled.Among all kinds of antidiabetic medications, metformin is recommended as the first-line antihyperglycemic management for type 2 diabetes. Insulin secretagogue,repaglinide is still one of the most widely used antidiabetic medications in China. However, there were few studies comparing the effects of these two medications on glycaemic control in Chinese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* All participants with type 2 diabetes, diagnosed by World Health Organization criteria, were recruited from outpatient of the Endocrinology Department in Shanghai Renji Hospital

Exclusion Criteria:

* Patients who had a history of coronary heart disease, abnormal renal function, active liver disease, chronic metabolic acidosis (including diabetic ketoacidosis), or severe chronic gastrointestinal disease.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline | week 12

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Renji Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai